CLINICAL TRIAL: NCT02359461
Title: Evaluation of the Effect of Pulsatile Cuts Stendo3 on Vascular Function Patients With Diabetes Type 2
Acronym: STENDO3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: STENDO, 17 rue du port 27400 LOUVIERS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CHU-0216
Record Dates: First submitted 2014-12-23; First posted 2015-02-10 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes
Keywords: Vascular function; Pulsatile cuts; Type 2 diabetes; Endothelium; Cardiovascular risk; Vasomotricity; FMD (Flow Mediated Dilatation)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Stendo group (Experimental): Subjects will be randomized into two groups determining the sequence: stendo then control, or control then stendo
  Interventions: Device: Combination pulsatile Stendo3
- control group (Other): Subjects will be randomized into two groups determining the sequence: stendo then control, or control then stendo
  Interventions: Device: Combination pulsatile Stendo3

INTERVENTIONS:
Device: Combination pulsatile Stendo3

SUMMARY:
The purpose of the study is to demonstrate an improvement of vascular function, and particularly dependent vasodilation flow and micro-vasculature, by STENDO for diabetic patients compared to a control period in crossover.

Action by shear stress causing vasodilation away from the microcirculation, STENDO should have a beneficial effect on vascular function in type 2 diabetics. These effects could be both treble just after the completion of a session with the device, and chronic with a potentiating effect of different sessions.

The investigators propose to study the different vascular function evaluation parameters we have, to highlight these acute and chronic changes. The investigators will also study the physical abilities to change topics and behavioral changes (spontaneous physical activity in particular) and impact on subject quality of life.

DETAILED DESCRIPTION:
Patients will be screened during a visit V0. A collection of consent (informed consent form), clinical examination and a fasting blood test will be carried out during this visit. Laboratory tests run-in will be composed of: Cell Blood Count (CBC) platelets, renal function tests (serum electrolytes, urea and creatinine), liver function tests, fasting blood glucose levels and Lipid Profile). Measurement of blood Pressure (2 successive measurements at intervals of 5 min) and an electrocardiogram will be realized. The different information collected at enrollment will allow stratification of cardiovascular risk by reference integrators scores (ESC-SCORE (European Society of Cardiology Score) and Framingham Heart Study).

The feasibility of measures for study criteria (functional measurements and assays) will be tested fasting during this visit as the blood test.

V0: Patient Pre-Inclusion: J-5 and J-10

* Patient Information
* Collection of informed consent
* Demographic data, weight / height, waist circumference
* Interrogation,
* Clinical examination, Electrocardiogram
* Measuring blood pressure (2 successive measurements at intervals of 5 minutes)
* ESC-SCORE (European Society of Cardiology Score) and Framingham Heart Study
* Criteria inclusion / non inclusion
* Functional Measurements (which will validate the feasibility on the patient)
* Blood test fasting: Complete Blood Count (CBC) platelets, renal function tests (serum electrolytes, urea, creatinine), liver function, and blood sugar, Lipid Profile.

V1 - Day 1 of the study At V1, patients have a clinical examination and a blood test fasting for the determination of endothelial parameters (Endothelial Micro Particles EMP).

Subjects will be randomized into two groups determining the sequence: STENDO then control, or control then STENDO .

Furthermore, the functional measurements will be performed at baseline, the morning after fasting for 12 hours in a room specially dedicated to the study of vascular reactivity (calm, stable temperature between 23 and 25 ° C).

When the patient has the STENDO technical, biological and functional assessments will be renewed at the end of the first session STENDO (immediately after).

* Clinical examination
* Confirmation of inclusion
* Allocation of randomization
* Measuring blood pressure (2 successive measurements at 5min interval)
* Blood Sample: Endothelial Micro Particles (EMP), Creatinine, Glucose, Glycated Haemoglobin (HbA1c), Lipid profile, Insulin
* Analysis of 24-hour urine: creatinine and microalbuminuria
* Functional Measures: Flow-mediated dilatation (FMD), Velocity time integral (VTI), Laser Doppler Flowmetry (LDF) , Stiffness of the central arteries by SphygmoCor , Stiffness of the central arteries and peripheral arteries by pOpmètre, fasting
* Measurements of physical abilities: endurance of the quadriceps and Maximum Voluntary Contraction (MVC), MVC hands, Aerobic capacity (VO2 max), 6 minutes Walk Test (6MWT), International Physical Activity Questionnary - French Version (IPAQ), Physical activity recorded by triaxial accelerometry (eMouve®),
* Measurement of quality of life : Visual Analogic Scale (VAS) and Short-form 36 Health survey (SF36).
* Stendo Session 1 hour or 1 hour rest according to the randomization group
* Blood Sample: Endothelial Micro Particles (EMP) (if STENDO)
* Realization of functional measures: FMD, VTI, FLD, SphygmoCor, pOpmètre, fasting after the 1st STENDO session (if STENDO)

For three months, patients will benefit from one-hour sessions of STENDO three times a week.

V2 30 days after inclusion +/- 1 week and V3 60 days after inclusion +/- 1 week - intermediate visits V2 and V3 intermediate visits will avoid lost sight especially during the monitoring period.

An evaluation of the quality of life (SF-36 and VAS) and physical activity (IPAQ questionnaire control and collection of eMouve) will be made for the 2 groups.

V4 at 90 days after inclusion +/- 1 week or End of 1st period V4 visit will take place in the same way that the V1 visit the day after the last session STENDO (where applicable): clinical examination, functional measurements, fasting blood test, measures of physical functions.

* Clinical examination
* Measuring blood pressure (2 successive measurements at 5min interval)
* Blood Sample: Endothelial Micro Particles (EMP), Creatinine, Glucose, Glycated Haemoglobin (HbA1c), Lipid profile analysis, Insulin
* Functional Measures: Flow-mediated dilatation (FMD), Velocity time integral (VTI), Laser Doppler Flowmetry (LDF) , Stiffness of the central arteries by SphygmoCor , Stiffness of the central arteries and peripheral arteries by pOpmètre, fasting
* Measurements of physical abilities: endurance of the quadriceps and Maximum Voluntary Contraction (MVC), MVC hands, Aerobic capacity (VO2 max), 6 minutes Walk Test (6MWT), International Physical Activity Questionnary - French Version (IPAQ), Physical activity recorded by triaxial accelerometry (eMouve®),
* Visual Analogic Scale (VAS) and Short-form 36 Health survey (SF36).

The time interval between V4 and V5 will be a minimum of 30 days to make a "wash-out" of stendo technique.

V5 : at least 120 days after inclusion, at least 30 days after "Wash-out" period Start of the 2nd period

V5 visit is the first visit of the second period of the crossover. This corresponds to the basal measurement of the second period.

The same assessments that will be carried out with V1 measuring parameters acute when the subject starts a period stendo

* Clinical examination
* Measuring blood pressure (2 successive measurements at 5min interval)
* Blood Sample: Endothelial Micro Particles (EMP), Creatinine, Glucose, Glycated Haemoglobin (HbA1c), Lipid profile analysis, Insulin
* Functional Measures: Flow-mediated dilatation (FMD), Velocity time integral (VTI), Laser Doppler Flowmetry (LDF) , SphygmoCor, pOpmètre, fasting
* Measurements of physical abilities: endurance of the quadriceps and Maximum Voluntary Contraction (MVC), MVC hands, Aerobic capacity (VO2 max), 6 Minutes Walk Test (6MWT), International Physical Activity Questionnary - French Version (IPAQ), Physical activity recorded by triaxial accelerometry (eMouve®),
* Visual Analogic Scale (VAS) and Short-form 36 Health survey (SF36).

If Stendo, for three months, patients will benefit from one-hour sessions of stendo three times a week.

V6 30 days +/- 1 week after the 2nd period onset and V7 60 days +/- 1 week after the 2nd period onset - intermediate visits The intermediate visits V6 and V7 will avoid lost sight especially during the monitoring period.

An evaluation of the Health-related quality of life by Visual Analogic Scale (VAS) and Short-form 36 Health survey (SF36)) and physical activity by International Physical Activity Questionnary - French Version (IPAQ) and Physical activity recorded by triaxial accelerometry (eMouve®) will be made for the 2 groups.

V8 90 days +/- 1 week End of second period Same measurements as the V4 visit. Signed by the investigator from the end of the study.

The day after the last session STENDO (where applicable): clinical examination, blood and functional measurements fasting blood test, physical function.

* Clinical examination
* Measuring blood pressure (2 successive measurements at 5min interval)
* Blood Sample: Endothelial Micro Particles (EMP), Creatinine, Glucose, Glycated Haemoglobin (HbA1c), Lipid profile analysis, Insulin
* Functional Measures: Flow-mediated dilatation (FMD), Velocity time integral (VTI), Laser Doppler Flowmetry (LDF) , SphygmoCor, pOpmètre, fasting
* Measurements of physical abilities: endurance of the quadriceps and Maximum Voluntary Contraction (MVC), MVC hands, Aerobic capacity (VO2 max), 6 Minutes Walk Test (6MWT), International Physical Activity Questionnary - French Version (IPAQ), Physical activity recorded by triaxial accelerometry (eMouve®),
* Visual Analogic Scale (VAS) and Short-form 36 Health survey (SF36).
* End of study forms

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Age between ≥ 18 and ≤ 75 years
* Diagnosis of diabetes> 2 years
* Asymptomatic on the cardiovascular
* No known heart disease
* ECG in sinus rythm with no signs suggestive of heart disease
* Absence of myocardial ischemia demonstrated by a stress test, myocardial scintigraphy or stress ultrasound
* Oral treatment with antidiabetic and / or insulin and / or incretin
* Affiliated with a social security scheme
* Having signed an informed consent

Exclusion Criteria:

* Type 1 diabetes
* Previous history of cardiomyopathy or ischemic heart disease
* Absence of sinus rythm
* ECG that suggest heart disease
* Electrical malfunction during the exercise test
* Hemo-dynamically significant valvular pathology
* Severe renal impairment (GFR <30 ml / min / 1.73m²)
* Uncontrolled hypertension: SBP ≥ 140 mm Hg or DBP ≥ 90 mm Hg The introduction or modification of antihypertensive treatment leads to the inability to include the subject for two months, the time to reach a new balance.
* Comorbidity involving life-threatening
* BMI> 40 kg /m2
* Peripheral vascular disease:
* Stage 3
* IPS (Index of systolic pressures) uninterpretable for which a doppler has diagnosed arteritis
* IPS lowered below 0.80
* Proximal or distal arterial bypass (or sub-popliteal fossa) or aortic prosthesis
* Deep vein thrombosis or superficial scalable recent lower limb or having a pulmonary embolism for less than one year
* Unhealed wound of the lower limbs or abdomen (ulcer, saphenectomy scars, surgical scarpa or abdominal approach)
* Disabling painful symptomatology of the lower extremities (paraesthesia, neuropathy, myalgia)
* Treaty by selective phosphodiesterase inhibitor (Sildenafil ...)
* Patients with cognitive impairment disabling

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in endothelial function of the large vessels by FMD (Flow Mediated Dilatation) | at baseline
  measured at baseline, then fasting at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study) separated by 1 month wash-out period

SECONDARY OUTCOMES:
Velocity of hyperemic response (VTI) | at day 1
Changes on Velocity of hyperemic response (VTI) | at baseline
  measured at baseline, then fasting at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Changes on circulating EMP levels (Endothelial MicroParticles) | at baseline
  measured at baseline, then fasting at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Stiffness of the central arteries by SphygmoCor | at day 1
Changes on Stiffness of the central arteries (SphygmoCor) | at baseline
  measured at baseline, then fasting at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Changes on Stiffness of the central arteries and peripheral arteries (finger / toe) (pOpmètre) | at baseline
Muscular Endurance quadriceps (in seconds) | at day 1
  measured at baseline, then fasting at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Changes on Maximal voluntary contraction quadriceps (MVC_q in Newton) | at visits just before and after 3 months
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Changes on Maximal voluntary contraction hand (MVC_h in Newton) | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Physical activity detected by a physical activity Questionnaire (IPAQ short) | at day 1
Changes on Aerobic capacity (VO2max) | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study)
Changes on 6-minute walk test (6MWT) | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment (Parallel part of the study)
Changes on Physical activity assessed by the International Physical Activity Questionnaire (IPAQ short) | at visits monthly during the 3 months of STENDO
  measured at visits monthly during the 3 months of STENDO (cross-over part of the study) and during the 3 months of control treatment (Parallel part of the study)
Changes on Physical activity recorded by triaxial accelerometry (eMouve®) | at visits monthly during the 3 months of STENDO
  measured at visits monthly during the 3 months of STENDO (cross-over part of the study) and during the 3 months of control treatment (Parallel part of the study)
Changes on Body composition (Fat mass, Muscle mass, Hydric mass) measured by impedancemetry | at visits measured at visits just before and after 3 months of STENDO
  measured at visits measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment ( Parallel part of the study)
Assessment of medications and posology | at visits monthly during the 3 months of STENDO
  measured at visits monthly during the 3 months of STENDO (cross-over part of the study) and during the 3 months of control treatment ( Parallel part of the study)
Changes on Health-related Quality of life assessed by the patient on a visual analogue scale (EVA_Quality of life) | at visits monthly during the 3 months of STENDO
  measured at visits monthly during the 3 months of STENDO (cross-over part of the study) and during the 3 months of control treatment ( Parallel part of the study)
Changes on Health related Quality of life according to the SF 36 Health survey assessed by patients | at visits monthly during the 3 months of STENDO
  measured at visits monthly during the 3 months of STENDO (cross-over part of the study) and during the 3 months of control treatment ( Parallel part of the study)
Changes on Health related quality of life using Visual analogue scale (VAS ) assessed by patients | at visits monthly during the 3 months of STENDO
  measured at visits monthly during the 3 months of STENDO (cross-over part of the study) and during the 3 months of control treatment (Parallel part of the study)
Changes on fasting Glycemia | at baseline
  measured at baseline, then fasting at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment ( Parallel part of the study)
Changes on Insulin serum levels | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment ( Parallel part of the study)
Changes on Glycated Haemoglobin serum levels (HbA1c) | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment ( Parallel part of the study)
Changes on Lipid profile on serum levels (total cholesterol, LDL / HDL, trigycérides) | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment ( Parallel part of the study)
Changes on Serum creatinine levels | at visits just before and after 3 months of STENDO
  measured at visits just before and after 3 months of STENDO (cross-over part of the study) and before and after 3 months of control treatment ( Parallel part of the study)
Assessment of Urinary creatinine levels | at day 1
Assessment of microalbuminuria levels of 24 hours | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Valensi P, Barber-Chamoux N, Rezki A, Lambert C, Pereira B, Duale C, Delmas D, Duclos M. Effects of single and multiple sessions of lower body diastole-synchronized compressions using a pulsating pneumatic suit on endothelium function and metabolic parameters in patients with type 2 diabetes: two controlled cross-over studies. Cardiovasc Diabetol. 2022 Dec 22;21(1):286. doi: 10.1186/s12933-022-01710-6. PMID 36550568